CLINICAL TRIAL: NCT05938634
Title: Efficacy of Stage Matched Intervention Based on the Transtheoretical Model of Change in Enhancing Female High School Students' Readiness to Engage in Regular Physical Exercise: A Randomized Controlled Trial
Brief Title: A Randomized Controlled Trial Using Stage-matched Intervention Based on the Transtheoretical Model of Change to Enhance Engaging in Regular Physical Exercise Among High School Female Students.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Collaborators: Nisreen Hameed Jebur (Unknown)
Responsible Party: Principal Investigator, Mohammed Baqer Habeeb Abd Ali, Faculty member, University of Baghdad
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: Regular Physical Exercise TTM
Record Dates: First submitted 2023-06-28; First posted 2023-07-10 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Physical Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants in the control group will be masked from the proposed intervention.
  Participants in the study group (in each Stage of Change) will be masked from the type of intervention they are supposed to receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Precontemplation (Experimental): The intervention that would involve the Processes of Change that people use when they would be in the Precontemplation Stage of Change.
  Interventions: Behavioral: Stage-matched interventions
- Contemplation-based intervention (Experimental): The intervention that would involve the Processes of Change that people use when they would be in the Contemplation Stage of Change.
  Interventions: Behavioral: Stage-matched interventions
- Preparation-based intervention (Experimental): The intervention that would involve the Processes of Change that people use when they would be in the Preparation Stage of Change.
  Interventions: Behavioral: Stage-matched interventions
- Action-based intervention (Experimental): The intervention that would involve the Processes of Change that people use when they would be in the Action Stage of Change.
  Interventions: Behavioral: Stage-matched interventions
- Maintenance-based intervention (Experimental): The intervention that would involve the Processes of Change that people use when they would be in the Maintenance Stage of Change.
  Interventions: Behavioral: Stage-matched interventions

INTERVENTIONS:
Behavioral: Stage-matched interventions — Precontemplation-based intervention Contemplation-based intervention Preparation-based intervention Action-based intervention Maintenance-based intervention

SUMMARY:
A randomized controlled trial that uses a Stage-matched intervention based on the Transtheoretical Model of Change to enhance engaging in regular physical exercise among high school female students.

DETAILED DESCRIPTION:
A randomized controlled trial that uses a Stage-matched intervention based on the Transtheoretical Model of Change to enhance engaging in regular physical exercise among high school female students.

The researchers will use two groups (study and control) in which participants will be randomly selected and assigned in each of the study and control groups using simple random sampling.

The study intervention will be designed based on each Stage of Change of the Transtheoretical Model of Change in that participants in each Stage of Change will receive the intervention that matches the Stage of Change they would be in.

A 12-week interval would be considered between administering the intervention and posttest 1 and the same interval would be used between posttest 1 and posttest 2.

ELIGIBILITY:
Inclusion Criteria:

* High school female students who do not experience any physical disability.

Exclusion Criteria:

* High school female students who experience any physical disability.

Ages: 15 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — High school female students
Enrollment: 144 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Engaging in regular physical exercise | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided